CLINICAL TRIAL: NCT01436175
Title: A Phase 3, Open-label, Multicenter, 12-month Extension Safety and Tolerability Study of SPD489 in Combination With an Antidepressant in the Treatment of Adults With Major Depressive Disorder With Residual Symptoms or Inadequate Response Following Treatment With an Antidepressant
Brief Title: SPD489 Adult Major Depressive Disorder (MDD) Open-label Safety and Tolerability Rollover Extension Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: SPD489 failed to demonstrate a benefit as adjunctive treatment to antidepressants. Termination was not related to any new safety findings.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD489-329; 2011-003019-47 (EudraCT Number)
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Lisdexamfetamine Dimesylate; Antidepressive Agents

ARMS (1):
- SPD489 + Antidepressant (Experimental)
  Interventions: Drug: SPD489 (Lisdexamfetamine dimesylate) + Antidepressant

INTERVENTIONS:
Drug: SPD489 (Lisdexamfetamine dimesylate) + Antidepressant — SPD489 20mg, 30mg, 50mg, or 70mg + Antidepressant (either escitalopram oxalate, sertraline hydrochloride, venlafaxine hydrochloride extended release or duloxetine hydrochloride) oral, once daily for 52 weeks
  Other Names: Vyvanse, LDX

SUMMARY:
This study is an optional continuation of previous short-term adult major depressive disorder (MDD) augmentation studies. Patients may only take part in this long-term, open-label research study if they completed a previous double-blind MDD augmentation study using SPD489.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed 1 of the respective short-term antecedent SPD489 MDD studies and did not experience any clinically significant AEs in the antecedent study that would preclude exposure to SPD489.

Exclusion Criteria:

* Subject has any current co-morbid Axis I or Axis II psychiatric disorder (including a lifetime history of psychosis) which was not present or recognized at entry into the antecedent study or has a concurrent chronic or acute illness or unstable medical condition that may deteriorate that could confound the results of safety assessments, increase risk to the subject or lead to difficulty complying with the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1570 (Actual)
Dates: Start 2012-02-27 (Actual); Primary Completion 2014-03-27 (Actual); Study Completion 2014-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (212):
- United States (140):
  - Birmingham Research Group, Birmingham, Alabama
  - ResearchOne, Inc., Scottsdale, Arizona
  - Arkansas Psychiatric Clinical Research Trials, P.A., Little Rock, Arkansas
  - South Coast Clinical Trials, Inc., Anaheim, California
  - American Neuropsychiatric Research, Inc., Carson, California
  - Catalina Research Institute, LLC, Chino, California
  - Shanti Clinical Trials, Colton, California
  - ATP Clinical Research, Costa Mesa, California
  - Clinical Innovation, Inc., Costa Mesa, California
  - Diligent Clinical Trials, Downey, California
  - Synergy Clinical Research Center of Escondido, Escondido, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - UC, Irvine Child Development Center, Irvine, California
  - Irvine Center For Clinical Research, Irvine, California
  - Omega Clinical Trials, LLC, La Habra, California
  - Semel Institute for Neuroscience & Human Behavior at UCLA, Los Angeles, California
  - Pacific Research Partners, Oakland, California
  - North County Clinical Research, Oceanside, California
  - Pasadena Research Institute, LLC, Pasadena, California
  - Anderson Clinical Research, Redlands, California
  - BreakThrough Clinical Trials, LLC, San Bernardino, California
  - Affiliated Research Institute, San Diego, California
  - PCSD - Feighner Research, San Diego, California
  - Clinical Innovations, Inc., San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Neuropsychiatric Center of Orange County, Santa Ana, California
  - Caliifornia Neuroscience Research Medical Group, Sherman Oaks, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Western Affiliated Research Institute, Denver, Colorado
  - Connecticut Clinical Research, Cromwell, Connecticut
  - Geriatric and Adult Psychiatry, LLC, Hamden, Connecticut
  - Institute of Living - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - CNS Clinical Research Group, Coral Springs, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Emerald Coast Mood & Memory, PA, Fort Walton Beach, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Amit Vijapura MD, Jacksonville, Florida
  - Psychiatric Associates, Lake City, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Fidelity Clinical Research Inc, North Miami, Florida
  - Scientific Clinical Research Inc., North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Compass Research, LLC, Orlando, Florida
  - Ali A. Kashfi, MD, PA, Orlando, Florida
  - Meridien Research, St. Petersburg, Florida
  - Comprehensive Clinical Development, Inc., St. Petersburg, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Kolin Research Group, Winter Park, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Atlanta Institute of Medicine & Research, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Institute for Behavioral Medicine, LLC, Smyrna, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - American Medical Research, Inc., Oakbrook Terrace, Illinois
  - Psyichiatric Medicine Associates, LLC, Skokie, Illinois
  - Sleep and Behavior Medicine Institute, Vernon Hills, Illinois
  - Davis Clinic, Indianapolis, Indiana
  - Pedia Research, LLC, Newburgh, Indiana
  - Northwest Indiana Center for Clinical Research, Valparaiso, Indiana
  - Clinical Trials Technology, Inc., Prairie Village, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - MCM Clinical Research LLC, Florence, Kentucky
  - Pedia Research, LLC, Owensboro, Kentucky
  - Louisiana Clinical Research LLC, Shreveport, Louisiana
  - Pharmasite Research, Inc., Baltimore, Maryland
  - Potomac Grove Clinical Research Center, Gaithersburg, Maryland
  - Office of Marc Hertzman, MD, Rockville, Maryland
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - Comprehensive Psyichatric Associates, Gladstone, Missouri
  - The Center for Pharmaceutical Research PC, Kansas City, Missouri
  - Private Practice - Howard J. Ilivicky, O'Fallon, Missouri
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Mid-America Clinical Research, St Louis, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Premier Psychiatric Research Institute, Lincoln, Nebraska
  - Clinical Research Consortium, Las Vegas, Nevada
  - Center For Emotional Fitness, Cherry Hill, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - CRI Worldwide, LLC, Willingboro, New Jersey
  - Albuquerque Neuroscience Inc., Albuquerque, New Mexico
  - Brooklyn Medical Institutes, Brooklyn, New York
  - Comprehensive Clinical Development, Inc., Fresh Meadows, New York
  - Bioscience Research LLC, Mount Kisco, New York
  - Clinilabs, Inc., New York, New York
  - Medical & Behavioral Health Research, PC, New York, New York
  - Fieve Clinical Research, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Montefiore Medical Center, The Bronx, New York
  - Sleep Medicine Centers of Western New York, West Seneca, New York
  - Triangle Neuropsyhiatry, Durham, North Carolina
  - Clinical Trials of America, Hickory, North Carolina
  - Dr. Richard Weisler, Raleigh, North Carolina
  - Northcoast Clinical Trials, Beachwood, Ohio
  - Community Research, Inc., Cincinnati, Ohio
  - Ohio State University Department of Psychiatry, Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Lindner Center for Hope, Mason, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - SP Research, PPC dba Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon) Inc., Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Paramount Clinical Research, Bridgeville, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Belmont Center for Comprehensive Treatment, Philadelphia, Pennsylvania
  - CRI Worldwide LLC, Philadelphia, Pennsylvania
  - UPMC Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - University Services, West Chester, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Medical University of South Carolina, Anxiety Disorders Program, North Charleston, South Carolina
  - Psychiatric Consultants, PC, Franklin, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - FutureSearch Clinical Trials, LP, Austin, Texas
  - KRK Medical Research, Dallas, Texas
  - Future Search Trials of Dallas, LP, Dallas, Texas
  - Pillar Clinical Research, LLC, Dallas, Texas
  - Bay Area Clinical Services, Friendswood, Texas
  - Houston Clinical Trials, LLC, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Wharton Research Center, Inc., Wharton, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Ericksen Research and Development, Clinton, Utah
  - Alliance Research Group, Richmond, Virginia
  - Summit Research Network (Seattle) LLC, Seattle, Washington
  - Dean Foundation for Health, Research, and Education, Middleton, Wisconsin
  - Independent Physician Consultants (dba IPC Research), Waukesha, Wisconsin
- Canada (14):
  - Dr. Alexander McIntyre Inc, Penticton, British Columbia
  - Dr. D. McIntosh & Dr. K. Kjernisted Clinical Research Inc., Vancouver, British Columbia
  - Chatham-Kent Clinical Trials Research Centre, Chatham, Ontario
  - Anxiety and Mood Disorder Center, Mississauga, Ontario
  - Dr. Sunny Johnson Medical Corporation, Medican Research Associates, Mississauga, Ontario
  - A. K. Karan Holdings, Ltd., Oakville, Ontario
  - International Sleep Clinic, West Parry Sound Health Centre, Parry Sound, Ontario
  - START Clinic for Mood and Anxiety Disorders, Toronto, Ontario
  - Sleep & Alertness Clinic, Toronto, Ontario
  - Manna Research, Toronto, Ontario
  - Recherches Neuro-Hippocampe, Gatineau, Quebec
  - l'Hopital Louis H. Lafontaine, Montreal, Quebec
  - Kells Medical Research Group Inc., Pointe-Claire, Quebec
  - Q & T Research Sherbrooke Inc., Sherbrooke, Quebec
- Chile (4):
  - Especialidades Medicas L y S, Las Condes, Santiagio
  - Centro de Estudios Clinicos (CEC), Providencia, Santiago Metropolitan
  - Biomedica Research Group, Providencia, Santiego
  - Psicomed Estudio Medicos, Antofagasta
- Czechia (9):
  - Psychiatrie Ricany, Říčany, Praha Vychod
  - Saint Anne s.r.o., Psychiatricka ambulance, Brno
  - Psychiatricka ambulance, Brno
  - Medicana s.r.o., Hořovice
  - Supervize s.r.o., Kutná Hora
  - Bialbi s.r.o., Litoměřice
  - Clintrial s.r.o., Prague
  - Psychiatry Trial, s.r.o, Prague
  - Medical Services Prague s.r.o., Prague
- Estonia (4):
  - Marienthal Psychiatry & Psychology Center of Mustamae, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Jaanson & Laane Ou, Tartu
  - Tartu University Hospital, Tartu
- Finland (3):
  - ARTES Psykiatrinen Palvelukeskus Oy, Helsinki
  - Satucon Oy / Privater, Kuopio
  - Puutonin Psykiatripalvelu, Turku
- Germany (10):
  - Facharzt fur Neurologie und Psychiatrie, Berlin
  - Emovis GmbH, Berlin
  - Complete Facharzt fur Neurologie und Psychiatrie, Berlin
  - Private Practice Drs. Bitter/Schumann, Bochum
  - ZSL Zentrum fuer medizinische Studien in Leipzig, Leipzig
  - Complete Karlstr, München
  - Studienzentrum Klinikum Nuernberg, Nuremberg
  - Somni bene GmbH, Schwerin
  - Gemeinschaftspraxis fur Neurologie und Psychiatrie, Westerstede
  - Medizinisches Studienzentrum Wuerzburg, Würzburg
- Hungary (2):
  - Semmelweis Egyetem Pszichiatrial es Pszichoterapias Klinkia, Budapest
  - Debreceni Egyetem Orvos es Egeszsegtudomanyi Centrum, Debrecen
- Mexico (2):
  - B&B Investigaciones Medicas, SC, Sinaloa, Mazatian
  - CRI Centro Regiomontano de Investigacion Clinica S.C, Nuevo León, Monterrey
- Poland (9):
  - Prywatne Gabinety Lekarskie "Promedicus" Anna Agnieszka Tomczak, Bialystok
  - Zespol Opleki Zdrowotnej w Chelmole, Chełmno
  - Centrum Badan Klinicznych PI-House sp. z o. o., Gdansk
  - Centrum Badan Klinicznych Pl-House, Gdansk
  - Klinika Chorob Psychicznych i Zaburzen Nerwicowych Uniwersyteckie Centrum Kliniczne, Gdansk
  - Klinika Chorob Psychicznych i Zaburzen Nerwicowych, Gdansk
  - Centrum Psychiatrii i Psychoterapi, Gorlice
  - NZOZ Syntonia, Kielce
  - Samodzieiny Publiczny Zespol Zakladow Opieki Zdrowotnej w Zurominie, Żuromin
- Puerto Rico (2):
  - Dharma Institute and Research Center, San Juan
  - INSPIRA Clinical Research, San Juan
- Romania (3):
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Alexandru Obregia" Sectia Clinica Psihiatrie I, Bucharest
  - Lorentina 2102 SRL, Târgovişte
  - Spitalui Clinic Judetean Mures, Târgu Mureş
- South Africa (3):
  - Cape Trial Centre, Bellville, Cape Town
  - Somerset West Clinical Research Unit, Somerset West, Western Cape
  - Flexivest Fourteen Research Centre, Cape Town
- Spain (7):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Fundacion de Alcorcon, Madrid
  - Centro de Salud Mental II la Corredoria, Oviedo
  - Centro de Salud Alamedilla Unidad de Salud Mental, Salamanca
  - Complejo hospitalario de Zamora, Zamora
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrolled eligible adults with major depressive disorder (MDD) who had completed treatment in a short-term antecedent SPD489 (lisdexamfetamine dimesylate) MDD study (SPD489-209 [NCT01435759], SPD489-322 [NCT01436149], and SPD489-323 [NCT01436162]).
Groups:
- SPD489 + Antidepressant: SPD489 20, 30, 50 or 70 milligram (mg) once daily orally for 52 weeks along with the assigned background product that participant had received during the antecedent study (antidepressant: either escitalopram oxalate, sertraline hydrochloride [HCl], venlafaxine HCl extended-release, or duloxetine HCl) at a dose consistent with applicable local labeling guidelines.
Period: Overall Study
Arm/Group | SPD489 + Antidepressant
Started | 1570
Completed | 300
Not Completed | 1270
Not completed — Adverse Event | 111
Not completed — Protocol Violation | 49
Not completed — Withdrawal by Subject | 108
Not completed — Lost to Follow-up | 89
Not completed — Lack of Efficacy | 24
Not completed — Met blood pressure or pulse withdrawal | 63
Not completed — Other | 826

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who took at least 1 dose of investigational product and had at least 1 post-Visit 0 (Week 0) safety assessment in this study.
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1559
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (11.89)
Age, Customized [Count of Participants; unit: Participants]
  18-55 Years | 1333
  56-65 Years | 226
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1056
  Male | 503
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1190
  Estonia | 24
  Hungary | 4
  Czech Republic | 83
  Mexico | 27
  Canada | 36
  Finland | 8
  Spain | 6
  Poland | 20
  Romania | 8
  South Africa | 5
  Chile | 33
  Germany | 69
  Argentina | 27
  Australia | 13
  United Kingdom | 1
  Croatia | 5

OUTCOME MEASURES:

1. Primary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviour during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behaviour occurred. The assessment is done by the nature of the responses, not by a numbered scale.
Time Frame: Week 5 up to Week 52/Early Termination(ET)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1559
participants
  Positive Suicidal Ideation | 68
  Suicidal Attempt | 4

2. Primary Outcome: Change From Baseline in Systolic Blood Pressure at Week 52
Description: Baseline was defined as the Augmentation Baseline Visit of the antecedent study (SPD489-209 [NCT01435759], SPD489-322 [NCT01436149], and SPD489-323 [NCT01436162]).
Time Frame: Baseline, Week 52/ET
Population: Safety Analysis Set. Here n = participants evaluable at specified time-points.
Measure: Mean (Standard Deviation); unit: millimeter of mercury(mmHg)
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1559
millimeter of mercury(mmHg)
  Baseline (n = 1559) | 117.6 (11.13)
  Change at Week 52/ET (n = 1558) | 2.4 (10.37)

3. Primary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 52
Description: as for outcome 2
Time Frame: Baseline, Week 52/ET
Population: Safety Analysis Set. Here n = participants evaluable at specified time-points.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1559
mmHg
  Baseline (n = 1559) | 75.4 (8.15)
  Change at Week 52/ET (n = 1558) | 1.2 (7.94)

4. Primary Outcome: Change From Baseline in Pulse Rate at Week 52
Description: as for outcome 2
Time Frame: Baseline, Week 52/ET
Population: Safety Analysis Set. Here n = participants evaluable at specified time-points.
Measure: Mean (Standard Deviation); unit: beats per minute(bpm)
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1559
beats per minute(bpm)
  Baseline (n = 1559) | 72.7 (9.90)
  Change at Week 52/ET (n = 1558) | 5.2 (10.58)

5. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 52/ET
Description: Designed to evaluate the extent to which illness symptoms impact a participant's life in 3 areas: work, social, and family/home. Each area is scored on a scale from 0 (no impairment) to 10 (highly impaired) with a total score ranging from 0 (unimpaired) to 30 (highly impaired). Lower scores translate into less impairment. Baseline was defined as the Augmentation Baseline Visit of the antecedent study (SPD489-209 [NCT01435759], SPD489-322 [NCT01436149], and SPD489-323 [NCT01436162]).
Time Frame: Baseline, Week 52/ET
Population: Full Analysis Set (FAS) included all participants in the Safety Analysis Set who had at least 1 clinical experience outcome assessment in the study. Here n = participants evaluable at specified time-points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1556
units on a scale
  Baseline (n=1548) | 12.7 (7.06)
  Change at Week 52/ET (n = 1530) | -4.3 (7.77)

6. Secondary Outcome: Number of Participants With Improvement on Clinical Global Impressions - Global Improvement (CGI-I)
Description: Participants who did not have Clinical Global Impressions - Severity of Illness (CGI-S) assessed at Week 8 in the antecedent study should not have had CGI-I assessed in this study and were excluded from the summary of CGI-I. CGI-I consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement includes a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: Week 52/ET
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1345
participants | 1021

7. Secondary Outcome: Short Form-12 Health Survey Version 2 (SF-12V2)
Description: SF-12V2 is a multi-purpose, 7-item survey that measures 8 domains of health: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. It is expressed by two summary measures (Aggregate Physical and Aggregate Mental) for which values can range from 0 to 100. A higher score is indicative of a better health state.
Time Frame: Week 52/ET
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1531
units on a scale
  Aggregate Physical | 49.1 (9.67)
  Aggregate Mental | 42.7 (11.55)

8. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self Report Questionnaire (EQ-5D-5L): Mobility
Description: Quality of life was assessed using the EQ-5D-5L, which is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is represented by a single item with 5 levels of responses
Time Frame: Week 52/ET
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1537
participants
  No problems in walking about | 1193
  Slight problems in walking about | 237
  Moderate problems in walking about | 82
  Severe problems in walking about | 24
  Unable to walk about | 1

9. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self Report Questionnaire (EQ-5D-5L): Self-Care
Description: as for outcome 8
Time Frame: Week 52/ET
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1537
participants
  No problems washing or dressing myself | 1304
  Slight problems washing or dressing myself | 174
  Moderate problems washing or dressing myself | 49
  Severe problems washing or dressing myself | 9
  Unable to wash or dress myself | 1

10. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self Report Questionnaire (EQ-5D-5L): Usual Activities
Description: as for outcome 8
Time Frame: Week 52/ET
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1537
participants
  No problems doing my usual activities | 800
  Slight problems doing my usual activities | 475
  Moderate problems doing my usual activities | 197
  Severe problems doing my usual activities | 55
  Unable to do my usual activities | 10

11. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self Report Questionnaire (EQ-5D-5L): Pain/Discomfort
Description: as for outcome 8
Time Frame: Week 52/ET
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1537
participants
  No pain or discomfort | 715
  Slight pain or discomfort | 536
  Moderate pain or discomfort | 208
  Severe pain or discomfort | 68
  Extreme pain or discomfort | 10

12. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self Report Questionnaire (EQ-5D-5L): Anxiety/Depression
Description: as for outcome 8
Time Frame: Week 52/ET
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1537
participants
  Not anxious or depressed | 461
  Slightly anxious or depressed | 687
  Moderately anxious or depressed | 289
  Severely anxious or depressed | 73
  Extremely anxious or depressed | 27

13. Secondary Outcome: EuroQoL Group 5-Dimension 5-Level Self Report Questionnaire (EQ-5D-5L): Visual Analog Scale
Description: EQ-5D-5L is one of the most widely used generic index measures of health-related quality of life. EQ-5D-5L Visual Analog Scale score is numbered from 0 to 100, where a score of 100 is the best health a participant can imagine
Time Frame: Week 52/ET
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1537
units on a scale | 75.7 (18.35)

14. Secondary Outcome: Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR)
Description: QIDS-SR is a validated, self-reported rating scale that contains 16 items scored on a scale from 0-3 with total scores ranging from 0 (no depression) to 27 (very severe depression). Lower scores indicate less depression. The QIDS-SR was only assessed in the SPD489-322 antecedent study. The QIDS-SR total score is calculated as the sum of the highest score on any 1 of Items 1-4, Item 5, the highest score on any 1 of Items 6-9, Items 10-14, the highest score on either Item 15 or 16.
Time Frame: Week 52/ET
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 506
units on a scale | 6.9 (4.48)

15. Secondary Outcome: Quality of Life Enjoyment Satisfaction Questionnaire Short Form (Q-LES-Q-SF)
Description: The Q-LES-Q-SF is a 16-item self-report questionnaire which evaluates general participant satisfaction with health, mood, relationships, functioning in daily life, and their treatment. Each item is rated on a 5-point scale from 1 (very poor) to 5 (very good). The total raw score (summary scale score) was calculated by summing item scores 1 to 14 (total raw score range: 14 to 70). Item 15 (satisfaction with medication, raw score range: 1 to 5) and Item 16 (overall satisfaction and contentment; raw score range: 1 to 5) were stand-alone items. For reporting, summary scale, Item 15 and Item 16 raw scores were transformed into percentage maximum possible score which ranged from 0 to 100, where higher scores are indicative of greater enjoyment or satisfaction.
Time Frame: Week 52/ET
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure, n = participants evaluable for specified categories
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 506
units on a scale
  Summary Scale (n = 506) | 61.5 (17.22)
  Satisfaction with Medication (n = 478) | 68.6 (19.66)
  Overall Satisfaction and Contentment (n = 506) | 63.2 (21.58)

16. Secondary Outcome: Change From Baseline in Sexual Functioning Questionnaire - 14 Item Scale (CSFQ-14) Total Score at Week 52/ET
Description: CSFQ-14 is a 14 item self-report tool that evaluates sexual functioning. Each item is scored on a 5-point Likert scale ranging from 1 (never) to 5 (always) with total scores ranging from 14 to 70. Higher scores reflect better sexual functioning. Baseline was defined as the Augmentation Baseline Visit of the antecedent study (SPD489-209 [NCT01435759], SPD489-322 [NCT01436149], and SPD489-323 [NCT01436162]).
Time Frame: Baseline, Week 52/ET
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 508
units on a scale
  Male: Baseline (n=167) | 46.6 (9.17)
  Male: Change at Week 52/ET (n=164) | 1.7 (7.16)
  Female: Baseline (n=341) | 37.2 (9.65)
  Female: Change at Week 52/ET (n=330) | 2.8 (8.33)

17. Secondary Outcome: Amphetamine Cessation Symptom Assessment (ACSA) Total Score
Description: ACSA scale has 16 symptom items rated on a scale from 0 (not at all) to 4 (extremely) with a possible total score range of 0 to 64. Higher scores indicate greater withdrawal symptom severity.
Time Frame: Week 53
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 1349
units on a scale | 14.3 (10.59)

18. Secondary Outcome: Patient Resource Utilization Questionnaire - Major Depressive Disorder (PRUQ-MDD)
Description: The PRUQ-MDD assessed the long term economic outcomes. It collects utilization of healthcare resources reported by the study participants. Participants answered the following questions: 1. Were you hospitalized in the past month, 2. Do you work for pay, 3. If you missed time at work last week, please note all the reasons why, 4. Would you say that the past week was typical, like the rest of the 3 weeks this month, in terms of your working hours, 5. Do you do volunteer work (VW), and 6. If you do not receive money for your work and do not participate in volunteer work, the reason is. Number of participants with response is reported.
Time Frame: Week 52/ET
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure
Measure: Number; unit: participants
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 482
participants
  Hospitalized in Past Month | 4
  Work for Pay | 337
  Reason Missing Work Time: Had a Day Off | 24
  Reason Missing Work Time: Physically Ill | 10
  Reason Missing Work Time: Upset/Depressed/Nervous | 15
  Reason Missing Work Time: Other | 36
  Past Week Was Typical: Yes | 249
  Past Week Was Typical: No, Worked More Hours | 43
  Past Week Was Typical: No, Worked Less Hours | 45
  Volunteer Work | 86
  Reason no Money/VW: Physically Ill | 6
  Reason no Money/VW: Upset/Depressed/Nervous | 30
  Reason no Money/VW: Cannot Find Work | 39
  Reason no Money/VW: Other | 48
  Reason no Money/VW: Not Applicable | 348

19. Secondary Outcome: PRUQ-MDD - Number of Days of Resource Utilization
Description: The PRUQ-MDD assessed the long term economic outcomes. It collects utilization of healthcare resources reported by the study participants. Number of nights in medical/surgical ward, number of nights in ICU, and number of days a participant received home care in the past month are reported.
Time Frame: Week 52/ET
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: days
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 482
days
  Number of nights in medical/surgical ward (n=4) | 1.3 (0.50)
  Number of nights in ICU (n=4) | 0.0 (0.00)
  Number of days received home care in past month | 0.0 (0.00)

20. Secondary Outcome: PRUQ-MDD - Number of Events (Visit to Health Care Provider/Visit to Hospital Facilities/Number of Times a Test Was Performed)
Description: The PRUQ-MDD assessed the long term economic outcomes. It collects utilization of healthcare resources reported by the study participants. Participants answered following questions - 1. How many times did you visit the following healthcare providers in the past month: Family doctor/primary care, Non-physician healthcare practitioner (NPHP), Psychiatrist/Psychologist/Counselor (PPC); 2. How many times did you take one of the tests, mentioned below, during the past month: Blood test, CT Scan, X Ray, Renal function, Thyroid function; and 3. How many times did you visit the hospital emergency room (ER), urgent care facility (UCF) or an after-hours clinic (AHC) in the past month. Number of events (visit to health care provider, visit to hospital facilities, and number of times a test was performed) are reported.
Time Frame: Week 52/ET
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: events
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 482
events
  Visit to Family doctor/primary care (n=481) | 0.2 (0.58)
  Visit to NPHP(n=480) | 0.1 (0.43)
  Visit to PPC(n=481) | 0.1 (0.86)
  Test performed: Blood Test (n=480) | 0.2 (2.30)
  Test performed: CT Scan (n=480) | 0.0 (0.08)
  Test performed: X Ray (n=480) | 0.0 (0.20)
  Test performed: Renal function (n=480) | 0.0 (0.00)
  Test performed: Thyroid function (n=480) | 0.0 (0.09)
  Test performed: Other test (n=479) | 0.1 (0.49)
  Visit to Hospital ER, UCF or AHC (n=482) | 0.0 (0.23)

21. Secondary Outcome: PRUQ-MDD - Number of Hours
Description: The PRUQ-MDD assessed the long term economic outcomes. It collects utilization of healthcare resources reported by the study participants. Participants answered following questions - 1. How many hours do you usually work or would you usually be expected to work (hrs/week); 2. How many hours did you actually work last week; 3. On average, how many hours do you volunteer per week. Number of hours are reported.
Time Frame: Week 52/ET
Population: FAS. Here, Number of Participants Analyzed = participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 482
hours
  Work or usually expect to work (n=337) | 34.0 (11.85)
  Actual work (n=337) | 31.2 (15.13)
  Average volunteer per week (n=86) | 8.6 (8.94)

22. Secondary Outcome: PRUQ-MDD - Effect of Depressive Symptoms
Description: The PRUQ-MDD assessed the long term economic outcomes. It collects utilization of healthcare resources reported by the study participants. Participants answered following questions on a 0 to 10 point scale - 1. During past week, how much did depressive symptoms affect work productivity; 2. During past week, how much did depressive symptoms affect regular non-work daily activities. Higher scores indicates more effect of depressive symptoms on work productivity and non-work daily activities.
Time Frame: Week 52/ET
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | SPD489 + Antidepressant
Number analyzed (Participants) | 482
units on scale
  Affected work productivity (n= 335) | 2.1 (2.37)
  Affected regular non work daily activities (n=482) | 2.5 (2.43)

ADVERSE EVENTS:
Time Frame: Up to Week 53
Description: Treatment-Emergent Adverse Events (TEAEs) were defined as Adverse Events (AEs) that started or deteriorated on or after the date of the first dose of investigational product and no later than 3 days after the last dose of investigational product.
Arm/Group | SPD489 + Antidepressant
Serious Adverse Events (participants affected / at risk) | 33/1559
Other Adverse Events (participants affected / at risk) | 921/1559
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD489 + Antidepressant (N=1559)
Angina pectoris (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Intestinal strangulation (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Non-Cardiac chest pain (General disorders) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Depressive symptom (Psychiatric disorders) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 3 (3)
Suicide attempt (Psychiatric disorders) | 3 (3)
Renal cyst (Renal and urinary disorders) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD489 + Antidepressant (N=1559)
Dry mouth (Gastrointestinal disorders) | 212 (233)
Nausea (Gastrointestinal disorders) | 116 (132)
Fatigue (General disorders) | 80 (82)
Feeling jittery (General disorders) | 82 (89)
Irritability (General disorders) | 79 (87)
Nasopharyngitis (Infections and infestations) | 137 (156)
Upper respiratory tract infection (Infections and infestations) | 100 (117)
Decreased appetite (Metabolism and nutrition disorders) | 189 (210)
Dizziness (Nervous system disorders) | 91 (102)
Headache (Nervous system disorders) | 241 (347)
Anxiety (Psychiatric disorders) | 83 (94)
Bruxism (Psychiatric disorders) | 89 (97)
Insomnia (Psychiatric disorders) | 204 (235)

LIMITATIONS AND CAVEATS:
The study was terminated on 11 Feb 2014. SPD489 failed to demonstrate a benefit as adjunctive treatment to antidepressants. Termination was not related to any new safety findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multi-centre publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multi-centre Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.